CLINICAL TRIAL: NCT07312201
Title: Oral Nutritional Supplementation in Children With Growth Concerns: A Randomized, Controlled Single-blinded Study
Brief Title: Oral Nutritional Supplementation in Children With Growth Concerns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2304INF
Record Dates: First submitted 2025-01-07; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Growth; Toddlers; Attention; Cognitive Function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Oral Nutritional Supplement (ONS) with Dietary Counselling (Experimental): The ONS is a nutrient dense oral nutritional supplement provided in powdered form, coupled with dietary counselling conducted by a trained dietitian over a 24-week period.
  Interventions: Dietary Supplement: Nutrient dense oral nutritional supplement
- Control: Dietary Counselling (No Intervention): Dietary counselling conducted by a trained dietitian over a 24-week period

INTERVENTIONS:
Dietary Supplement: Nutrient dense oral nutritional supplement — The ONS is provided in powdered form that provides the appropriate amount of protein, vitamins and minerals
  Arms: Experimental: Oral Nutritional Supplement (ONS) with Dietary Counselling

SUMMARY:
Multi-center, single-blinded, randomized, controlled study consisting of two arms, to investigate the impact of an oral nutritional supplement in combination with dietary counseling on growth in children with growth concerns as compared to children who receive dietary counselling alone

ELIGIBILITY:
Inclusion Criteria:

* Child's parent(s) is of legal age of majority (18 years of age), must understand the informed consent form and other relevant study documents, and is willing and able to fulfill the requirements of the study protocol.
* Evidence of a personally signed and dated informed consent document indicating that the child's parent(s) / legally acceptable representative (LAR) has been informed of all pertinent aspects of the study.
* Child was full-term at birth (i.e., ≥ 37 completed weeks of gestation with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg).
* Child is aged 24 - 41 months at inclusion.
* Child is generally healthy (acute illnesses in a minor condition which are common in childhood such as viral or bacterial infections (e.g., conjunctivitis, otitis media, upper/lower respiratory tract infection, gastroenteritis, hand foot & mouth disease) at time of enrolment is permitted).
* Children whose parents, caregivers, or guardians show some concern about their child's dietary intakes and growth, such as child is too thin for his or her height, or child has experienced recent rapid weight loss or failure to gain weight or height and child has a z-score for weight-for-age or weight-for-height or both parameters ≤ -1SD as per WHO growth charts.
* Child's parents agree to feed their child an oral nutritional supplement in addition to normal diet.
* Child's parent(s) / guardian can be contacted directly by telephone throughout the study.

Exclusion Criteria:

* Child is currently breastfed or is consuming breast milk.
* Child is currently consuming or consumed in the past month growing-up milk / toddler formula. Growing-up milks / toddler formulas are products specifically formulated for young children and provide key macro- and micro-nutrients.
* Child is currently consuming or consumed in the past month oral nutrition supplement (ONS). The standard ONS formula has an energy density of at least 0.85 kcal/mL, containing protein, carbohydrate and/or fat, as well as a wide range of micronutrients to supplement or use as the sole source of nutrition.
* Child has known or suspected cows' milk protein intolerance / allergy, lactose intolerance, galactosemia, soy intolerance / allergy, fish oil intolerance / allergy, or allergy or intolerance to any ingredient in the study product.
* Child fed vegan, vegetarian, or vegetarian plus fish diets in which milk products are excluded.
* Underlying medical illness that could affect growth or feeding, such as gastrointestinal [GI] disorders (such as celiac disease, short bowel syndrome, maldigestion/malabsorption, significant GI malformations or surgery etc.); neurodevelopmental disability; chronic infections (such as tuberculosis or HIV infection); congenital disease or genetic disorders (such as congenital cardiac disease, Down syndrome, thalassemia); or other chronic illness that may impact growth or feeding according to the clinician opinion.
* Child is unable to consume foods or ONS orally (e.g. dysphagia, anorexia, difficulty in swallowing due to acquired or congenital abnormalities that would hamper oral intake of the study product.)
* Clinically significant nutritional deficiency requiring specific nutritional therapy other than the study product (for example tube feeding)
* Child has acute illness including acute viral infection, respiratory tract infection etc. even in a minor condition at time of enrolment. A child presenting with an acute illness can be re-screened at least two weeks after the episode of illness has resolved.
* Child has a z-score for weight-for-height or weight-for-age or height-for-age or any combination of these three parameters ≤ -3SD as per WHO growth charts.
* Children currently receiving or having received prior to enrolment medication which are known to impact growth including systemic steroids, growth hormone and insulin
* Child or child's parent(s) not willing and/or not able to comply with scheduled visits and/or have plans to relocate to a different geographical location from the study location during the study period.
* Child of any investigational site staff member or Nestlé employee directly involved in the conduct of the trial.
* Child is currently participating in or has participated in another clinical trial within 4 weeks prior to enrolment.

Ages: 24 Months to 41 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2026-09-30 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of ONS coupled with dietary counseling on growth in children | Day 1 to Day 169
  Change in weight-for-age z score

SECONDARY OUTCOMES:
Weight of growing children | Day -7 to Day 169
  Measurement of weight will be in grams
Length/height of growing children | Day -7 to Day 169
  Measurement of length/height will be in centimetres (cms)
Mid-upper arm circumference of growing children | Day -7 to Day 169
  Measurement of mid-upper arm circumference will be in centimetres (cms)
Body mass index (BMI) of growing children | Day -7 to Day 169
  Calculated BMI will be in kilograms per square metre (kg/m²)
Z-scores and percentiles | Day -7 to Day 169
  Change from baseline in sex-age-specific percentiles and z-scores
Nutrient intake of children | Day 1 to Day 169
  Paper-based 24-hour dietary recall administered by a trained dietitian on-site
Bone mass index of children | Day 1 to Day 169
  Bone density will be measured in z-scores
Physical strength of children | Day 1 to Day 169
  The grip strength will be measured in kilograms (kg)
Skeletal muscle mass of children | Day 1 to Day 169
  Urine sample will be collected in millimetres during the study (mL)
Blood marker of longitudinal growth | Day 1 to Day 169
  Blood sample will be collected during the study in microlitres (μL)
Blood markers of bone turnover | Day 1 to Day 169
  Blood sample will be collected during the study in microlitres (μL)
Blood markers of nutritional status | Day 1 to Day 169
  Blood sample will be collected during the study in microlitres (μL)
Cognitive Functioning | Day 169
  Questionnaire will be administered by the site staff for assessment
Product satisfaction of children and parents | Day 14 to Day 169
  Questionnaire will be administered by the site staff for assessment
Parental perceptions on appetite, growth, level of activity and sleep of children | Day 1 to Day 169
  Questionnaire will be administered by site staff for assessment
Safety assessment (Adverse Events) | Day -7 to Day 169
Duration of illness and absence from pre-school due to illness | Time Frame: Day -7 to Day 169
Concomitant medications and treatments | Day -7 to Day 169

IPD SHARING:
Plan to Share IPD: Undecided